CLINICAL TRIAL: NCT01819714
Title: Evaluation of the Impact of Care Based on Sensory Support for Elderly Patients Suffering From Alzheimer'S-type Neurodegenerative Disease
Brief Title: Sensory Support Care for Elderly Patients Suffering From Alzheimer'S-type Neurodegenerative Disease
Acronym: SensiCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PHRIP/2012/JD; 2013-A00005-40 (Other: RCB number)
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Alzheimer Disease
Keywords: Snoezelen; Multi-sensorial care session; Alzheimer's-type neurodegenerative disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study population (Experimental): Patients hospitalized at the Serre-Cavalier centre and who have Alzheimer's-type neurodegenerative disease (see inclusion criteria).
  Interventions: Other: Multi-sensory supportive care

INTERVENTIONS:
Other: Multi-sensory supportive care — The Serre-Cavalier center will implement Snoezelen-type multisensory care sessions for included patients; these care sessions correspond with the patients' daily hygiene/toilette care.
  The impact of this multisensory strategy will be evaluated using a before-after design.
  Other Names: Snoezelen-type care; Snoezelen toilette

SUMMARY:
The main objective of this study is to evaluate the effect of 3 months of "Snoezelen-type" multi-sensory care sessions on NeuroPsychiatric Inventory Questionnaire (NPI-Q) scores for patients with Alzheimer's-type neurodegenerative disease.

DETAILED DESCRIPTION:
The secondary objectives of this study are to study the following elements in relationship to the implementation of a "Snoezelen-type" multi-sensory care strategy for patients with Alzheimer's-type neurodegenerative disease:

A. to evaluate the effects on NPI-Q scores at 1 month, 6 months and 12 months .

B. evaluate the effects on quality of life (questionnaire QOL-AD) at 0 and 12 months.

C. assess changes in the "aggressive behavior" subsection of the Cohen-Mansfield Agitation Inventory (CMAI) questionnaire over 0, 1, 3, 6 and 12 months.

D. assess changes in drug consumption (anxiolytics, antidepressants, hypnotics, neuroleptics)over the study period

ELIGIBILITY:
Inclusion Criteria:

* The patient's legal representative must have given his/her informed and signed consent (or the patient if he/she is judged competent)
* The patient must be insured or beneficiary of a health insurance plan
* Alzheimer's-type neurodegenerative pathology
* The patient has been living in the participating center for > 2 months

Exclusion Criteria:

* The patient's legal representative refuses to sign the consent (or the patient if he/she is judged competent)
* It is impossible to correctly inform the patient's legal representative
* The patient has already has Snoezelen-therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in NPI-Q scores | 3 months

SECONDARY OUTCOMES:
Change from baseline in NPI-Q scores | 1 month
Change from baseline in NPI-Q scores | 6 months
Change from baseline in NPI-Q scores | 12 months
Change from baseline in the Quality-of-life-Alzheimer's Disease questionnaire (QOL-AD) | 12 months
Change from baseline in the "aggressive behavior" subsection of the Cohen-Mansfield Agitation Inventory (CMAI) questionnaire | 1 month
Change from baseline in the "aggressive behavior" subsection of the Cohen-Mansfield Agitation Inventory (CMAI) questionnaire | 3 months
Change from baseline in the "aggressive behavior" subsection of the Cohen-Mansfield Agitation Inventory (CMAI) questionnaire | 6 months
Change from baseline in the "aggressive behavior" subsection of the Cohen-Mansfield Agitation Inventory (CMAI) questionnaire | 12 months
Change in drug consumption from baseline | 1 month
Change in drug consumption from baseline | 3 months
Change in drug consumption from baseline | 6 months
Change in drug consumption from baseline | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jane Debuysschere, IDE, Study Director — Centre Hospitalier Universitaire de Nîmes; Jean-Marie Cros, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Centre de Gérontologie de Serre Cavalier, Nîmes, France